CLINICAL TRIAL: NCT00688298
Title: A Prospective, Single-Arm, Post Market Clinical Study to Evaluate a Mid-Urethral Vaginal Tape Procedure With a Pre-Pubic Delivery Approach, for the Treatment of Stress Urinary Incontinence
Brief Title: Post Market Clinical Study to Evaluate a Mid-Urethral Vaginal Tape Procedure With a Pre-Pubic Delivery Approach, for the Treatment of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Kurt Douglass, Boston Scientific
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0299
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2008-05

CONDITIONS: Stress Urinary Incontinence; Intrinsic Sphincter Deficiency
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (1):
- Arm 1 (Experimental): Female patients Greater than or 18 years of age, diagnosed with Stress Urinary Incontinence (SUI).
  Interventions: Device: Prefyx PPS™ System; Device: Advantage ™ System

INTERVENTIONS:
Device: Prefyx PPS™ System — A mesh implant intended for use as a suburethral sling for the treatment of stress urinary incontinence resulting from hypermobility and/or intrinsic sphincter deficiency.
Device: Advantage ™ System — The Advantage Mesh implant is intended as a suburethral sling for the treatment of stress urinary incontinence resulting from hypermobility and/or intrinsic sphincter deficiency.

SUMMARY:
The pre-pubic approach of the tension free vaginal sling placement is a new approach in the treatment of SUI. The retropubic approach of the tension free vaginal sling is the standard method of device delivery; in addition a suprapubic and a transobturator approach are alternative methods of delivery. All of these delivery approach systems are intended to place the mesh "tension free" in the mid-urethra.

There are currently no studies that investigate the pre-pubic delivery approach in the United States. However, the largest series of cases in Europe using the pre-pubic system was done by Ulmsten (published in the European Journal of Obstetrics and Gynecology and Reproductive Biology) 107 (2003) 205-207, titled " Pre-Pubic tension free vaginal tape application: an alternative to classic tension free vaginal tape application in selected patients with SUI."

The primary objective of this study is to evaluate the feasibility of using a pre-pubic approach to the placement of a mid-urethral vaginal mesh.

* Demonstrate the mesh can be properly placed in the mid-urethra using a pre-pubic approach;
* Assess the performance of the delivery device by measuring the ease of use, technical complexity, and instrument difficulties

ELIGIBILITY:
Inclusion Criteria:

* Female greater than 18 years of age
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Diagnosed with genuine SUI confirmed by urodynamic evaluation (urodynamic evaluations performed in the past 6 months are acceptable) and documented in the source documents as in patients charts, physicians notes, nurses notes, hospital records, etc.
* If the patient has an overactive bladder, the condition must be a minor component of the patient's disorder demonstrated by the urodynamic testing. This is a physician
* discretion for inclusion or exclusion in the study.
* Patients are willing to complete (PFDI-short form 20) and PISQ-12 at baseline, 3 months, 6 months and 12 months post-operatively.
* Patient has documented SUI classification and the degree of hypermobility and/ or intrinsic sphincter abnormality (Q-Tip test). Confirm the patient's SUI diagnosis using one or more of the following procedures:

  * Vaginal exam
  * Cough provocation test
  * Cystoscopic exam
* Patients must have a negative urine culture
* Patients' bladder capacity of 350cc or more
* Document voiding diary pre- and post-operatively
* Document post-void residual (PVR) of equal to or less than 100cc
* Patients that require a regional, general anesthesia or monitored anesthesia
* Pad test on baseline that demonstrate 5 grams or greater urine loss
* Patients are mentally competent and able to understand all study requirements
* Patients agree to read and sign the informed consent form prior to any study related procedures (screening/ baseline visit)

Exclusion Criteria:

* Patients who, in the clinical judgment of the investigator, are not suitable for this study
* Patients who, are in the investigator's opinion, mentally or legally incapacitated, or unable to read or understand written material, thereby preventing informed consent
* Patients who have participated in an investigational study (medical device or drug) within 30 days of study entry that may impact analysis of this device or have previously participated in the current trial
* Patients who are pregnant, lactating, or planning future pregnancies
* Patients with Diabetes Mellitus type I or II
* Patients with vesicourethral reflex, upper urinary tract obstruction, spastic bladder, or detrouser muscle instability
* Patient treated with corticosteriod or immunosuppresant agents within 90 days pre-operatively except for patients treated with inhaled steroids for the treatment of asthma
* Patients with compromised immune systems
* Patients with any acute cystitis or urethritis
* Patients that had previous urinary incontinence procedures
* Patients that had a previous radiation to the pelvis
* Patients with coagulopathy and/ or currently on anticoagulant medications
* Patients with known or suspected hypersensitivity to the mesh
* Patients that complain of pelvic pain and/ or dyspareunia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-05; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Measuring the amount of time to complete successful pre-pubic delivery approach and placement of the mesh in the mid-urethra and the number of difficulties associated with the placement | post procedure
Document all types and number of complications associated with the pre-pubic delivery approach and mesh placement in the mid-urethra | post procedure
Physician-Procedure satisfaction questionnaire | post procedure

SECONDARY OUTCOMES:
The percentage of patients who remain continent or improved following treatment at timed intervals | 10 days, 3 months, 6 months, 12 months
The percentage of patients who report substantial improvement and consider the surgery successful, as measured by patient self-reporting | 10 days, 3 months, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walsh, M.D., Study Director — Boston Scientific Corporation
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States